CLINICAL TRIAL: NCT06488287
Title: The Use of Transcranial Direct Current Stimulation (tDCS) to Reduce Emotional Eating in Tier 3 Obese Patients: A Randomised Controlled Feasibility Trial Protocol
Brief Title: tDCS and Emotional Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23039
Record Dates: First submitted 2024-05-07; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorders
Keywords: obesity; emotional eating; brain stimulation; tDCS
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity; Emotional Eating | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real stimulation (Experimental): Participants in this arm will receive 6 sessions of real tDCS.
  Interventions: Device: Transcranial direct current stimulation (brain stimulation)
- Sham stimulation (Placebo Comparator): Participants in this arm will receive 6 sessions of sham tDCS.
  Interventions: Device: sham Transcranial direct current stimulation (brain stimulation)

INTERVENTIONS:
Device: Transcranial direct current stimulation (brain stimulation) — The intervention will be applied using two sponge electrodes soaked in a saline solution. The stimulation montage will comprise left DLPFC anodal or sham stimulation. The reference (cathodal) electrode will be placed over the right supraorbital ridge, and the anodal electrode will be placed over the region corresponding to the left DLPFC (F3 of the EEG10-20 international system). The 2mA continuous current will be applied during the active stimulation condition via gradual ramps that start and stop after 30 seconds of stimulation (current ramps). For sham stimulation, the electrodes will remain in place for the whole session, but the current will only be applied for the first 36 seconds of the stimulation. Each tDCS session will last for 20 minutes.
  Arms: Real stimulation
Device: sham Transcranial direct current stimulation (brain stimulation) — The intervention will be applied using two sponge electrodes soaked in a saline solution. The stimulation montage will comprise left DLPFC anodal or sham stimulation. The reference (cathodal) electrode will be placed over the right supraorbital ridge, and the anodal electrode will be placed over the region corresponding to the left DLPFC (F3 of the EEG10-20 international system). For sham stimulation, the electrodes will remain in place for the whole session, but the current will only be applied for the first 36 seconds of the stimulation. Each tDCS session will last for 20 minutes.
  Arms: Sham stimulation

SUMMARY:
This research investigates the feasibility of undertaking a large, randomised control trial of transcranial direct current stimulation (tDCS) as a treatment modality for managing food cravings and emotional eating. This study explores how tDCS, a non-invasive brain stimulation technique, can influence brain activity and potentially impact appetite regulation, self-control, reward processing, and other factors related to weight management.

All participants will receive 6 sessions of stimulation within three weeks. the investigators aim to implement a two-day interval between intervention sessions, providing participants with a two-day rest period between sessions. This scheduling approach is intended to mitigate potential side effects and promote participants' recovery.

DETAILED DESCRIPTION:
Participants were invited to take part in this study based on their registration in the tier 3 bariatric service at the Royal Derby Hospital and a score of more than 6 in the binge eating survey previously completed as part of their clinical care. the invistigators invite 30-40 participants to participate in this study.

After the completion of the consent form participants will be asked to complete a safety questionnaire to check whether there are any known reasons tDCS would not be suitable for them. If it is suitable to participate in a tDCS study for obesity, participants will be randomised to either real tDCS or Sham tDCS (Sham tDCS is like a "fake" version of tDCS. It's used in experiments to make people think they're getting brain stimulation when they're not. This helps researchers see if the real brain stimulation has a genuine effect or if it's just because people believe it will work). The randomization process for group assignment will be conducted using a computer program, which means participants will not have the ability to select or choose their preferred group. participants will receive 6 sessions of real tDCS or sham for three weeks (2 sessions a week). the investigators will follow up with participants for two weeks after the study end. The follow-up procedure will involve the completion of questionnaires and the stop signal task once again. Additionally, body weight measurements will be taken during this stage. Therefore, they will participate for 8 weeks in this study. All sessions will take place in the University of Nottingham medical school at Derby Royal Hospital and University of Nottingham jubilee campus. The first and last session will take approximately 1.30 hours and the other sessions will last 40 minutes each. In the first and last sessions, participants will be asked to fill in 4 questionnaires (30 minutes to fill), doing an impulsivity test (also known as Stop Signal Task) (it is an easy test and will take 5 minutes. The stop signal task is a psychological test that measures participant ability to stop or pause a planned action when they're signalled to do so. It helps assess self-control and how well participants can inhibit or control their impulses) and receive one session of tDCS or sham (20 minutes). In the 4 sessions, the participant will only receive one session of real tDCS or sham. During the study (8 weeks) the participant will be asked to fill a daily food record using mobile app. After the end of the study, the participant will be asked to do an interview to talk about the experience of being in the study. The interview will be conducted at the end of the study either in person or online using Teams.

tDCS has no major safety concerns according to National Institute for health and Care Excellence (NICE 2015). The most frequent temporary side effects are mild tingling, slight itching, moderate fatigue, headache or, less frequently, a slight burning feeling. These effects usually develop at the start of the tDCS and disappear shortly after. Headaches, mild discomfort, or irritation on the skin generally involve slight discomforts that are promptly relieved by over-the-counter pain relief medicines. It is important to inform us of any side effects experienced after the tDCS sessions and to contact participant's GP or treating clinician with any healthcare concerns or study-related questions.

the investigators cannot promise the study will help the participant but the information that investigators get from this study may help to the advancement of scientific knowledge by expanding our understanding of the effects of tDCS on appetite regulation, cognitive control, and long-term behaviour modification in the context of obesity, potentially leading to the development of more effective treatments and interventions for weight management in the future.

the recruitment started on 01/03/2024 and the study end date will be 30/09/2025. this study was funded py the PGR office at the University of Nottingham.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity in tier 3.
* Capacity to consent to participate in research.
* Adults aged 18 to 65 years old.
* A high score in the emotional eating survey (minimum of 6 score in weight loss readiness questionnaire) (this will be taken from participant's medical note by usual care staff)

Exclusion Criteria:

* Non-obese patients (BMI<25).
* A history of epilepsy or other major neurological disorders
* Having pacemakers or other metal implants.
* No history of eating disorders or emotional eating.
* Pregnant patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Response rate and number of patients who met the inclusion criteria, agreed to participate in the study, and completed the study. | 5 weeks
  Response rate and number of patients who met the inclusion criteria, agreed to participate in the study, and completed the study.
Feasibility of completion study questionnaire. | 5 weeks
  number of patients who met the inclusion criteria, agreed to participate in the study, and completed the study questionnaire.
Means and standard deviations of scores on study questionnaires. | 5 weeks
  3. Means and standard deviations of scores on study questionnaires.
Dropout ratio in each group | 5 weeks
Safety of the intervention will be assessed by adverse event reported by patients | 5 weeks

SECONDARY OUTCOMES:
Body weight (Kg) | 5 weeks
BMI (kg/m^2) | 5 weeks
The Eating Disorder Examination Questionnaire (EDE-Q) | 5 weeks
  The Eating Disorder Examination Questionnaire (EDE-Q) is a widely used self-report measure for assessing the range and severity of eating disorder symptoms. It consists of 28 items and evaluates behaviours and attitudes associated with eating disorders over the past 28 days.
  The questionnaire is divided into four subscales: A global score of 2.3 is often used as a cut-off to identify probable eating disorders.
The Food Cravings Questionnaire-State (FCQ-S) | 5 weeks
  The Food Cravings Questionnaire-State (FCQ-S) measures momentary food cravings using a 15-item scale. Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). This gives the FCQ-S a minimum possible score of 15 and a maximum possible score of 75. High score means worse symptoms.
The Emotional Eating Scale II (EES-II) | 5 weeks
  The Emotional Eating Scale II (EES-II) is an extended version of the original Emotional Eating Scale (EES), designed to assess eating in response to both positive and negative emotions. The EES-II consists of 33 items, each rated on a 5-point scale from 0 (no desire to eat) to 4 (an overwhelming urge to eat). This results in a minimum score of 0 and a maximum score of 132.
  The EES-II includes subscales that measure eating in response to different emotional states:
  Anger/Frustration (9 items) Anxiety (8 items) Depression (10 items) Positive Emotions (6 items) Higher scores on the EES-II indicate a greater tendency to eat in response to emotional states, both positive and negative.
Calories consumption (using food record app) | 5 weeks
Impulsivity using stop signal task | 5 weeks
Adverse events | 5 weeks
The Food Craving Questionnaire-Trait (FCQ-T) | 5 weeks
  The Food Craving Questionnaire-Trait (FCQ-T) assesses the frequency and intensity of food cravings over time and consists of 39 items. Each item is rated on a 6-point Likert scale, where 1 indicates "never" and 6 indicates "always." The total score ranges from a minimum of 39 to a maximum of 234. Higher scores reflect greater food craving tendencies.
The Food Craving Inventory (FCI) | 5 weeks
  The Food Craving Inventory (FCI) is a self-report measure designed to assess the frequency of food cravings for specific food types over the past month. The FCI consists of 28 items, each rated on a 5-point scale from 1 (never) to 5 (always/almost every day). This gives the FCI a minimum possible score of 28 and a maximum possible score of 140. high score means worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Derby, Royal Derby Hospital Centre Uttoxeter Road, United Kingdom

IPD SHARING:
Plan to Share IPD: No